CLINICAL TRIAL: NCT07227688
Title: Evaluation of the Proximal Anatomical Form Quality of Different Precontoured Sectional Matrix Systems in Complex Proximal Posterior Resin Composite Restorations: Randomized Clinical Trial.
Brief Title: Evaluation of the Proximal Form of Precontoured Sectional Matrix in Complex Proximal Posterior Restorations
Acronym: RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona mahmoud Abd Elrahman, Lecturer, Conservative Dentistry Department, Faculty of Dentistry, Cairo University, Cairo, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mona_international_2
Record Dates: First submitted 2025-11-08; First posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Complex Caries
Keywords: proximal anatomical form; precontoured sectional matrix; complex restorations; Randomized Clinical Trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Sectional matrix: Classic ring system (Experimental): Sectional matrix: Classic ring system (TOR VM, Moscow, Russia)
  Interventions: Device: Sectional matrix: Classic ring system (TOR VM, Moscow, Russia)
- BioFit Posterior Matrix System (Active Comparator): BioFit Posterior Matrix System (Bioclear, Tacoma, Washington, USA).
  Interventions: Device: BioFit Posterior Matrix System
- Saddle system (Active Comparator): Saddle system (TOR VM, Moscow, Russia)
  Interventions: Device: Saddle system (TOR VM, Moscow, Russia)

INTERVENTIONS:
Device: BioFit Posterior Matrix System — precontoured sectional matrix system
  Arms: BioFit Posterior Matrix System
Device: Saddle system (TOR VM, Moscow, Russia) — precontoured sectional matrix systems
  Arms: Saddle system
Device: Sectional matrix: Classic ring system (TOR VM, Moscow, Russia) — precontoured sectional matrix systems
  Arms: Sectional matrix: Classic ring system

SUMMARY:
Evaluation of the proximal anatomical form quality of different precontoured sectional matrix systems in complex proximal posterior resin composite restorations using Fédération Dentaire Internationale' (FDI) clinical criteria for the evaluation of direct and indirect restorations

DETAILED DESCRIPTION:
The importance of the interdental anatomy of a class II direct composite restoration is one of the most underestimated topics in direct posterior composite restorations. The proximal emergence profile of the restoration and the contact area should be designed to maximize arch continuity and to minimize food impaction. A thorough knowledge of proper contacts and contours and how they ought to be duplicated as well as predisposing factors for proximal contact loss as proximal caries, embrasure size and position, and marginal ridge location and thickness, all of which contribute to achieving ideal occlusal harmony.

Conventional circumferential matrix systems produced poor proximal contact points with proximal overhangs or open contacts, and they failed to produce optimum contact points; thus, their usage should be prohibited.

It was found that, optimum contact points were highly associated with the sectional matrix system; there was a 70% lower risk for non- optimum contact points than the circumferential matrix system. Open and tight contacts were highly associated with the circumferential matrix system regardless of operator experience. Sectional matrix systems with separation rings should be implemented as the first choice in clinical decision making for proximal posterior restorations.

Although in vitro and in vivo studies showed that the use a contoured sectional metal matrix band with a separation rings results in optimum contact point and emergence profile, its use is technique sensitive due to rounded contours and thin thickness of matrices, which can cause a depression or bending in the matrix material during placement, rendering it unusable. Also, this matrix systems have shortcomings and does not give the expected result in all class II cavities. The variation in depth, width of the box, distance between the cervical cavity margin and the adjacent tooth requires customization of the interproximal space.

As the main objective is to recreate proximal contacts and contour that mimic the natural teeth making this area self-cleansable, preserving the periodontium, improving the restoration durability as well as maintaining the mesio-distal dimension of either dental arch. This mission is more complicated with badly broken-down teeth. By defining a badly destructed tooth we can say that it is a tooth that has lost a significant amount of tooth material which may be due to caries affection, fractures, or even extensive endo treatments. The result is that the remaining tooth structure becomes friable and weakened and presents a challenge during restoration due to increased distance between the cervical cavity margin and the adjacent tooth and the situation is more complicated if part of the buccal and lingual walls are missing making the ordinary sectional matrix liable to collapse after placing the separation rings.

classic ring system made by TOR VM was chosen as the comparator. Several innovative types of sectional matrix systems were introduced to the market with several thicknesses, heights, profiles of curvature, variation of wedges and separation clamps. These advancements have enabled dentists to create the most beneficial proximal contact surfaces and anatomically correct contours, both of which are critical for tooth periodontal complex protection.

In badly broken-down teeth, the sectional matrix should have a correct curved profile, making it possible to create a correct emergence profile in a cervico-occlusal direction. An increased proximal curvature (cervico-incisally) of the matrix band is required when the distance between the cervical cavity margin and the adjacent tooth increases. This is observed when the cervical cavity margin is in a more apical position. Thus, to select the correct matrix band, one must be aware of its maximum curvature. Besides the matrix bands should have enough extensions in a buccolingual direction to be able to restore the contact area efficiently.

Hard stainless steel sectional saddle matrices (TOR VM, Moscow, Russia) have a maximum curvature of ±0.7 mm compared to ±0.5 mm of the classical TORVM sectional matrix. The maximum curvature starts more cervically, making it easier to reach deeper margins. And these matrices offer more buccal and lingual wrap than traditional matrices.

The Bioclear Biofit matrices introduce new matrix technology and designs that claimed by the manufacturer to ensure ideal proximal composite contour. BioFit Matrix bands (Bioclear Matrix Systems; Tacoma, WA, USA) have the highest maximum curvature among all available matrices in the market (±0.9 mm). These matrix bands are contoured plastic (Mylar) sectional matrices with a placement tab that makes the matrix easy to place. Transparent matrices may allow better light transmission and allegedly more effective polymerization of the underlying resin composite. Mylar matrices also leave the composite more polished and contoured than traditional metal matrices which leave a more matte finish. In addition, the new shape of the Biofit matrices offers 30% more buccal/lingual and occlusal wrap than traditional matrices and can be used in cavities that are more open in a bucco-lingual direction. In addition, the matrix features a curved occlusal embrasure, which, if the matrix is well-positioned, shortens the finishing time of the occlusal embrasure with burs or disks.

The clinical performance of these matrices regarding obtaining optimum contact, contour and prevents overhangs is yet to be evaluated. Controlled randomized clinical trials- based on correctly adopted evaluation systems, are crucial for effective evidence-based dental knowledge and restorative practice. Thus, this study aims to contribute in providing evidence-based literature concerning current innovative matrixing systems and an evidence based clinical practice in the most critical situation which is restoring contacts in badly broken down teeth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with posterior complex class II cavities to be restored with resin composite restorations.
* 18 - 45 years.
* Males or Females.
* Good oral hygiene.
* Co-operative patients approving to participate in the study.

Exclusion Criteria:

* Poor oral hygiene.
* Allergic history concerning methacrylates
* Evidence of parafunctional habits.
* Presence of malalignment of teeth

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a change in the proximal anatomical form using (FDI) World Dental Federation clinical criteria for the evaluation of direct and indirect restorations | Immediately after restoration placement at the baseline
  1. Proximal contact point with the aid of visual examination and 25-/50-/100-μm metal blades.
  2. Form and contour utilizing visual examination and radiographic assessment.
  For each criterion, one score will be chosen from 5 scores (excellent, good, satisfactory, unsatisfactory & poor).

CONTACTS AND LOCATIONS:
Overall Officials: Sherifa A Abd ElAziz, PhD, Study Director — Cairo University
Locations (1):
- Cairo University, Giza, GZ, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Markose, D. Restoring proximal contacts of teeth. IOSR J Dent Med Sci. 2017; 16: 46-9.
- [Background] Loomans BA, Opdam NJ, Roeters FJ, Bronkhorst EM, Burgersdijk RC, Dorfer CE. A randomized clinical trial on proximal contacts of posterior composites. J Dent. 2006 Apr;34(4):292-7. doi: 10.1016/j.jdent.2005.07.008. Epub 2005 Sep 12. PMID 16157438
- [Background] Hickel R, Roulet JF, Bayne S, Heintze SD, Mjor IA, Peters M, Rousson V, Randall R, Schmalz G, Tyas M, Vanherle G. Recommendations for conducting controlled clinical studies of dental restorative materials. Clin Oral Investig. 2007 Mar;11(1):5-33. doi: 10.1007/s00784-006-0095-7. Epub 2007 Jan 30. PMID 17262225
- [Background] Peumans M, Venuti P, Politano G, Van Meerbeek B. Effective Protocol for Daily High-quality Direct Posterior Composite Restorations. The Interdental Anatomy of the Class-2 Composite Restoration. J Adhes Dent. 2021;23(1):21-34. doi: 10.3290/j.jad.b916819. PMID 33512113
- [Background] Durr-E-Sadaf; Ahmad MZ, Gaikwad RN, Arjumand B. Comparison of two different matrix band systems in restoring two surface cavities in posterior teeth done by senior undergraduate students at Qassim University, Saudi Arabia: A randomized controlled clinical trial. Indian J Dent Res. 2018 Jul-Aug;29(4):459-464. doi: 10.4103/ijdr.IJDR_26_17. PMID 30127197
- [Background] Esteves H, Correia A, Araujo F. Classification of extensively damaged teeth to evaluate prognosis. J Can Dent Assoc. 2011;77:b105. PMID 21975072
- [Background] Shaalan, O. O., & Ibrahim, S. H. (2021). Clinical evaluation of sectional matrix versus circumferential matrix for reproduction of proximal contact by undergraduate students and postgraduate dentists: A randomized controlled trial. Journal of International Oral Health, 13(1), 10.